CLINICAL TRIAL: NCT03450213
Title: Comparison of Anterior and Posterior Corneal Astigmatism in Patients With Keratoconus and Controls
Brief Title: Astigmatism in Keratoconus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Mamdouh, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Keratoconus
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with keratoconus (Active Comparator): Pentacam will be used for comparison between astigmatism in patients with keratoconus and normal people at the same age and sex.
  Interventions: Device: Pentacam
- Normal people at the same age and sex (Placebo Comparator): Pentacam will be used for comparison between astigmatism in patients with keratoconus and normal people at the same age and sex.
  Interventions: Device: Pentacam

INTERVENTIONS:
Device: Pentacam — Pentacam will be used to measure the magnitude and axis orientation of anterior and posterior corneal astigmatism.

SUMMARY:
Keratoconus is a bilateral (but usually asymmetrical) non-inflammatory progressive thinning process of the cornea. It manifests as characteristic cone-like ectasia of the cornea associated with irregular stromal thinning, resulting in a cone-like bulge , which causing irregular astigmatism and vision impairment.

DETAILED DESCRIPTION:
Keratoconus is the most common form of corneal ectasia, with an incidence of 50-230 per 100,000 persons.Pentacam used diagnose & detect the progression in patients with keratoconus and also provide a detailed information about corneal tomography and topography.

In the last few years, it has been shown that in healthy individuals the posterior corneal surface has not only a different amount of astigmatism but also a different alignment of the steep meridian.

The aim of this research is to compare the amount and axis alignment of anterior and posterior corneal astigmatism in keratoconus with a healthy controlled group .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with keratoconus using the following criteria:

Specific diagnostic signs is asymmetric refractive errors with high progressive or irregular astigmatism, and elevated keratometry values, scissoring of the red reflex, Vogt striae, Fleischer rings, inferior or central steepening on topography with abnormal localized steepening .

Exclusion Criteria:

* Unwillingness to participate in the study .
* Corneal scarring.
* Any ectatic conditions that were not explicitly keratoconus such as keratoglobus and pellucid marginal degeneration .
* Previous ocular surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between astigmatism in patients with keratoconus and normal people. | Two years
  Pentacam will be used for comparison between astigmatism in patients with keratoconus and normal people at the same age and sex

REFERENCES:
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273